CLINICAL TRIAL: NCT06678048
Title: A Single-Arm, Two Stage, Phase II Study of Arsenous Acid Combined With Palliative Chemotherapy for Refractory Triple-Negative Breast Cancer
Brief Title: Arsenous Acid for Refractory Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-036
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — arsenous acid; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arsenous Acid plus Chemotherapy (Experimental): Arsenous Acid , Eribulin, Gemcitabine, Utidelone, Vinorelbine
  Interventions: Drug: Arsenous Acid plus Chemotherapy

INTERVENTIONS:
Drug: Arsenous Acid plus Chemotherapy — Arsenous Acid , Eribulin, Gemcitabine, Utidelone, Vinorelbine

SUMMARY:
The primary objective of this study is to assess the progression-free survival (PFS) and safety of arsenous acid in combination with palliative chemotherapy for refractory triple-negative breast cancer following multiple lines of treatment.

DETAILED DESCRIPTION:
The study is a Single-arm, two-stage, Phase II clinical trial. The main purposes of this study are to assess the efficacy and safety of arsenous acid in combination with palliative chemotherapy for refractory triple-negative breast cancer following multiple lines of treatment. Palliative chemotherapy regimen includes Eribulin, Gemcitabine, Utidelone and Vinorelbine, by the treatment of physician's choice (TPC). This study is designed based on Bayesian probability and divided into two stages. All patients will undergo tumor efficacy assessment every two cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Understands and voluntarily signs the informed consent form.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
* Life expectancy greater than 3 months
* Histologically or cytologically confirmed metastatic invasive breast cancer, with negative for hormone receptor (HR) and human epidermal growth factor receptor 2 (HER2). HR negative is defined as Immunohistochemistry (IHC) for estrogen receptor (ER) and/or progesterone receptor (PR) showing < 1% of tumor cells. HER2 negative is defined as IHC 0 or 1+, or IHC 2+ with a negative in-situ hybridization.
* Refractory to at least two prior standard therapeutic regimens for metastatic disease. For TNBC patients with a programmed death-ligand 1 (PD-L1/22C3) positive result (combined positive score, CPS ) ≥10, eligibility requires prior treatment with chemotherapy combined with PD-1. Additionally, TNBC patients with a known germline breast cancer susceptibility gene (BRCA) mutation, who are assessed to be unsuitable for or unable to receive poly (ADP-ribose) polymerase (PARP) inhibitor therapy by the physician, also qualify for the study. Recurrence within 12 months following TNBC adjuvant therapy is considered as first-line therapy.
* Eligible for one of the chemotherapy options listed as palliative chemotherapy (Eribulin, Gemcitabine, Utidelone, Vinorelbine) as per investigator assessment.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). At least one lesion must not have received prior radiotherapy and should qualify as a baseline lesion according to RECIST 1.1 criteria, with a measurable longest diameter of ≥10 mm on CT or MRI (for lymph nodes, the short axis must be ≥15 mm). Patients with only bone metastases are eligible for enrollment, as are patients with stable brain metastases.
* Patients must have adequate bone marrow reserves and normal organ function, as defined by the following criteria: Hemoglobin ≥ 9.0 g/dL. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L. Platelet count ≥ 100 × 10^9/L. Total bilirubin (TBL) ≤ 1.5 × upper limit of normal (ULN). Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN, except in cases of Hepatitis B Virus (HBV). For patients with liver metastases, ALT and AST ≤ 5 × ULN.
* Premenopausal women can use medically acceptable methods of contraception during the study.
* Demonstrates good compliance.

Exclusion Criteria:

* Uncontrolled hypertension, persistent or active infections.
* Persistent toxicities from prior antitumor treatments (excluding alopecia) that have not improved to Grade ≤ 2 or baseline levels, such as hearing loss, neuropathy, or immune-related toxicities (hypothyroidism/hyperthyroidism, hyperglycemia, adrenal insufficiency, etc.).
* Tumor-related spinal cord compression or active brain metastases.
* Significant third-space fluid retention (e.g., ascites or pleural effusion) deemed by the investigator to be unsuitable for study participation.
* Uncontrolled infections requiring intravenous antibiotics, antivirals, or antifungals.
* Participants known to be human immunodeficiency (HIV) positive, hepatitis B positive, or hepatitis C positive.
* Uncontrolled or significant cardiac disease, including myocardial infarction or unstable angina within the last six months, congestive heart failure, severe arrhythmias, or uncontrolled hypertension (resting systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg).
* Suspected interstitial lung disease (ILD) or non-infectious pneumonia that cannot be ruled out and requires corticosteroid treatment.
* Active autoimmune diseases or inflammatory conditions (including inflammatory bowel disease, systemic lupus erythematosus, sarcoidosis, granulomatosis with polyangiitis, rheumatoid arthritis, uveitis, autoimmune non-infectious pneumonia, and autoimmune myocarditis).
* Concurrent treatment with any other antitumor therapies.
* Subjects deemed unlikely to comply with the study procedures and requirements by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 10 months
  Progression-Free Survival (PFS) was defined as the time from enrollment until objective tumor progression by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No